CLINICAL TRIAL: NCT02866071
Title: Intranasal Ketamine as an Adjunct to Fentanyl for the Prehospital Treatment of Acute Traumatic Pain
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jason McMullan (Other)
Responsible Party: Sponsor-Investigator, Jason McMullan, Director, Fellowship in EMS Medicine; Director-Research, Division of EMS; Associate Professor of Emergency Medicine, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: McMullan Ketamine
Record Dates: First submitted 2016-08-05; First posted 2016-08-15 (Estimated); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Acute Traumatic Pain
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine (Active Comparator): 50mg IN Ketamine Hydrochloride
  Interventions: Drug: Ketamine Hydrochloride
- Placebo (Placebo Comparator): 50mg IN placebo
  Interventions: Drug: Placebo-Comparator

INTERVENTIONS:
Drug: Ketamine Hydrochloride — 50mg IN Ketamine Hydrochloride
  Arms: Ketamine
Drug: Placebo-Comparator — 50mg IN Placebo
  Arms: Placebo

SUMMARY:
STUDY SYNOPSIS Objectives The primary objective is to estimate the proportion of subjects who report clinically important reductions in pain score (defined as 2 points on a 0-10 verbal numerical rating scale) after receiving a single dose of fentanyl (per local standard) with or without intranasal (IN) ketamine (50mg) prior to hospital arrival for the treatment of acute traumatic pain.

Design and Outcomes This protocol describes two linked studies conducted as a prospective, randomized, placebo-controlled single-site clinical trial. The primary study has a primary outcome variable of reduction of reported pain of at least 2 points (on the 0-10 Verbal Numerical Rating Scale1,2) when comparing the pretreatment pain score to the pain score obtained upon reassessment 30 minutes after medication administration; secondary outcomes of the primary trial include reduction of reported pain at Emergency Department (ED) arrival; the incidence of adverse events; additional opiate requirements prior to ED arrival and in the first three hours of ED care. The secondary study explores secondary outcomes including: development of chronic pain (measured by the Brief Pain Inventory,3) or post-traumatic stress disorder (measured by the PTSD Checklist for DSM-54) and overall satisfaction with life (measured by the Satisfaction With Life Scale5) at 90-days after injury.

Interventions and Duration Adult men who qualify for prehospital pain treatment under paramedic standing orders will be screened for inclusion and will undergo informed consent for the primary trial. After ED arrival, subjects who consented for the primary trial will be approached for inclusion in the secondary trial. Prehospital consent for primary trial enrollment and study drug administration will occur concurrent with receiving a single dose of fentanyl (IV, IM or IN per current standard practice). Consenting subjects will be 1:1 randomized to receive either 50mg IN ketamine or IN saline placebo. Pain will be rated on a 0-10 scale by the subject prior to treatment and at 30 minutes following treatment and will receive further pain assessments at 30 minute intervals for the first three hours of their ED care. Additional pain medications given prior to hospital arrival and within the first three hours of ED care will also be recorded. The primary outcome of the primary trial will be reduction in baseline pain between the pretreatment measurement and 30 minutes after medication administration. Consent for the secondary trial will be obtained for the additional baseline assessments for secondary outcomes and at 90-day follow-up. Overall satisfaction with life and symptoms of PTSD and chronic pain will be assessed before hospital disposition (in-person) and via phone follow-up at 90-days (+/- 14 days) after injury.The subject will have the option to complete the 90-day follow-up assessments in-person if it coincides with a clinical appointment on the medical campus.

Sample size and Power We consider a 2-point reduction in pain to be clinically significant, and thus our primary outcome for the primary trial will compare the proportion of subjects achieving a 2-point reduction in pain at 30 minutes post-medication administration between the treatment group and the control group. Sample size considerations are based on this primary analysis. To test the hypothesis that the proportion of those treated with fentanyl alone that have at least a 2-point reduction in their pain will be lower than the proportion of those treated with the combination of fentanyl and single-dose ketamine who have a 2-point reduction in their pain, we will use a chi-square test (or the Fisher's Exact Test if appropriate). An intent to treat approach will be used. We expect the response rate in the two groups to be 40% and 60%, respectively. These estimates are based on the response rates in a study comparing pain management efficacy between subjects treated with morphine alone and morphine plus ketamine.6 With this magnitude of effect, a sample size of 97 per group will have 80% power to detect the difference between the two groups when the critical level of significance is set to 5%. To allow for subject drop-out, protocol deviations, and missing outcome data, we plan to enroll an additional 15% in each arm, for a total of 224 subjects.

ELIGIBILITY:
Adult males with acute traumatic pain that are eligible to receive pain medication prior to hospital arrival under current practice will be screened for enrollment in the primary trial. The inclusion and exclusion criteria mirror this existing protocol (Appendix 1: Prehospital Protocols).

Inclusion Criteria of Primary Trial

* Subjects must be experiencing pain due to acute trauma (i.e. extremity deformity, tourniquet placement, or severe burns).
* A Verbal Numerical Rating Scale pain score ≥7 prior to any pain medication administration.
* Age: ≥18 through 65 years (i.e. subjects must have had their 18th birthday, but not had their 66th birthday).
* Systolic blood pressure ≥100mmHg and <180mmHg.
* Transported directly from the scene of injury to the Emergency Department at University of Cincinnati Medical Center by a participating EMS agency.
* English-speaking.
* Male sex.
* Receiving fentanyl IV/IM/IN as part of standard care. Exclusion Criteria of Primary Trial
* Subject reported allergy to morphine, fentanyl, or ketamine.
* EMS treatment with ketamine (any), morphine (any), or more than one dose of fentanyl prior to enrollment.
* Inter-facility transfers.
* Prisoners or those in police custody.
* Female sex.
* Paramedic clinical concern of acute agitation or psychosis.
* Pain medication not needed in judgment of prehospital provider.
* Altered level of consciousness, mental status change, or suspected head injury.
* Paramedic clinical concern of circulatory shock.
* Inability to provide Verbal Numerical Rating Scale.
* Facial injury or suspicion of nasal bone fracture.
* Paramedic judgment that subject cannot consent due to underlying cognitive impairment.
* Systolic blood pressure ≥180mmHg

Justification for Exclusions Medications are generally withheld if there is a reported drug allergy. This is a study of acute pain management, and pretreatment with additional medications may bias results. EMS does not routinely provide inter-facility (between hospital) transfers, and these subjects will likely be transferred several hours after injury and should have received pain medications from the original hospital. Prisoners or those in police custody represent a protected population. Ketamine is pregnancy class N (unknown); while frequently used in developing countries for analgesia/sedation for Cesarean sections, 73-75 obtaining a serum or urine pregnancy test is not possible in the prehospital setting. Breast feeding women and women of childbearing age will be excluded. To avoid introducing bias from a partially included population, all women will be excluded. Ketamine may cause psychomotor agitation in some subjects (even though ketamine is frequently used as treatment of excited delirium76). Pre-existing agitation or mental status changes and inability to provide VNRS prevent outcomes assessments. Current prehospital protocols do not allow pain medications for patients with circulatory shock. Nasal trauma may interfere with medication delivery or absorption. Previous trials have excluded patients with a systolic blood pressure ≥180mmHg.6,38,49

Inclusion Criteria for Secondary Trial Subjects enrolled in the primary trial will be approached for participation in the secondary trial. Enrollment in the secondary trial will involve a second and separate consent process (further described below). Participation in the secondary trial is not required to participate in the primary trial.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2017-10-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in Pain | between pre-treatment EMS assessment (baseline) and at 30-minutes post-treatment
  reduction in reported pain of two or more points based on the Verbal Numerical Rating Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McMullan J, Droege C, Strilka R, Hart K, Lindsell C. Intranasal Ketamine as an Adjunct to Fentanyl for the Prehospital Treatment of Acute Traumatic Pain: Design and Rationale of a Randomized Controlled Trial. Prehosp Emerg Care. 2021 Jul-Aug;25(4):519-529. doi: 10.1080/10903127.2020.1808746. Epub 2020 Oct 15. PMID 32772873
- [Background] McMullan J, Droege C, Strilka CR, Lindsell C, Linke MJ. Food and Drug Administration and Institutional Review Board Approval of a Novel Prehospital Informed Consent Process for Emergency Research. Prehosp Emerg Care. 2021 Jul-Aug;25(4):512-518. doi: 10.1080/10903127.2020.1806969. Epub 2020 Sep 9. PMID 32790539
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873